CLINICAL TRIAL: NCT01800760
Title: Probiotics to Improve Women's Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Arkansas Children's Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 136010
Record Dates: First submitted 2013-01-28; First posted 2013-02-28 (Estimated); Last update posted 2023-12-20 (Actual); Status verified 2023-12

CONDITIONS: Healthy
Keywords: healthy; obese; women
MeSH Terms: conditions — Obesity | interventions — Probiotics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- No groups (Experimental)
  Interventions: Dietary Supplement: Probiotics

INTERVENTIONS:
Dietary Supplement: Probiotics — Probiotics once a day for three weeks.

SUMMARY:
The purpose of the study is explore the effect of probiotics on plasma lipopolysaccharides (LPS) concentrations, as well as insulin and glucose levels, in obese women prior to and after dietary challenges (high carbohydrate meal, high fat meal).

ELIGIBILITY:
Inclusion Criteria:

* BMI=30-40 kg/m2
* Healthy, age 18 or older
* Not consuming yogurt or cultured milk regularly (</= 1x/wk) or any probiotic supplement

Exclusion Criteria:

* Medical conditions or medications that may affect metabolism as determined by the PI.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2012-04 (Actual); Primary Completion 2019-05-20 (Actual); Study Completion 2019-05-20 (Actual)

PRIMARY OUTCOMES:
Plasma LPS concentrations | five weeks

SECONDARY OUTCOMES:
Glucose concentrations | five weeks

CONTACTS AND LOCATIONS:
Overall Officials: Aline Andres, PhD, Principal Investigator — University of Arkansas
Locations (1):
- Arkansas Children's Nutrition Center, Little Rock, Arkansas, United States